CLINICAL TRIAL: NCT02725983
Title: Psychological, Behavioral and Clinical Effects of Intra Oral Camera: a Randomized Control Trial on Adults With Gingivitis
Brief Title: Intra-oral Camera in Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Faculdade de Psicologia (Unknown)
Responsible Party: Principal Investigator, Mario Rui Araújo, Master in Health psychology, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06/2014
Record Dates: First submitted 2016-03-18; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Gingival Hemorrhage; Gingivitis; Health Behavior; Communication
Keywords: Gingivitis; Oral Hygiene; Intra oral camera; Self regulation; bleeding
MeSH Terms: conditions — Gingival Hemorrhage; Gingivitis; Health Behavior; Communication; Self-Control; Hemorrhage

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra Oral Camera (Experimental): Dental appointment, one hour and included activities that are normally part of a SPT consultation (Bardet et al. 1999), as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback as described by Newton and Asimakopoulou (2015). Special attention was given to patient communication and words such as 'cleaning' and 'hygiene' were replaced by therapeutic synonyms (e.g. inflamed areas and controlling the inflammation). In this group, the device SOPROCARE® by Acteon was used in the examination and diagnosis and also for the establishment of therapeutic goals, strategies and skills.
  Interventions: Behavioral: SPT consultation; Device: SOPROCARE®
- No Intra Oral camera (Active Comparator): Dental appointment, one hour and included activities that are normally part of a SPT consultation (Bardet et al. 1999), as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback as described by Newton and Asimakopoulou (2015) and considered crucial to the accomplishment of long term behavior change. Moreover, special attention was given to patient communication and words such as 'cleaning' and 'hygiene' were replaced by therapeutic synonyms (e.g. inflamed areas and controlling the inflammation) in order to focus patients´ attention on the varied facets of oral health care and increase their perception of the treatment needs. In this group, the device SOPROCARE® by Acteon was not used.
  Interventions: Behavioral: SPT consultation

INTERVENTIONS:
Behavioral: SPT consultation
Device: SOPROCARE®
  Arms: Intra Oral Camera

SUMMARY:
Evaluate the effects of using an intra-oral camera (IOC) during supportive periodontal therapy (SPT), on the psychological, behavioral and clinical parameters of patients with gingivitis, outlined by evidence and a theory-based framework.

DETAILED DESCRIPTION:
A group of 78 adult patients with gingivitis receiving an SPT was randomized into two groups: IOC and control.

Bleeding on Marginal Probing (BOMP), self-reported dental hygiene behaviors, and psychological determinants of behavior change (outcome expectancies, self-efficacy and planning) and IOC opinion were evaluated one week before or during the consultation and four months later.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old.
* + 20 teeth (minimum 5 per quadrant)
* BOMP > 0.5

Exclusion Criteria:

* periodontitis (pockets >4),
* smoking patients
* orthodontic patients
* pregnant
* 1 removable partial denture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The gingival condition was assessed using the BOMP (Bleeding on Marginal Probing) index , as described by Van der Weijden et al. (1994). | Baseline to 4 months
  In this index, bleeding is scored during 30 seconds of probing using a 3 point scale from 0 to 2 (0 - no bleeding, 1 - point bleeding, 2 - excess bleeding).

SECONDARY OUTCOMES:
Dental Hygiene (Flossing and tooth-brushing habits) | Baseline to 4 months
  In order to assess dental hygiene, two questions were asked on brushing and flossing habits. Individual scores for brushing and flossing were calculated and a composite score was also computed for both (referred to as Dental Hygiene). A 5 point Likert-scale was used. Item example: In the last two weeks/four months how often have you flossed your teeth?
Measuring Health Behavior Change: Health Action Process Approach Model (HAPA, Schwarzer, 2008) | Baseline to 4 months
  Measures adapted to oral health from previous studies with the HAPA model (Godinho et al. 2015) were used. All the psychological variables were evaluated using a 7 point Likert-type scale, ranging from totally disagree (1) to totally agree (7).

CONTACTS AND LOCATIONS:
Overall Officials: Maria-João Maria-João, PhD, Principal Investigator — Faculdade de Psicologia da Universidade de Lisboa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674
- [Background] Godinho CA, Alvarez MJ, Lima ML, Schwarzer R. Health messages to promote fruit and vegetable consumption at different stages: A match-mismatch design. Psychol Health. 2015;30(12):1410-32. doi: 10.1080/08870446.2015.1054827. Epub 2015 Jul 24. PMID 26010304
- [Background] Bardet P, Suvan J, Lang NP. Clinical effects of root instrumentation using conventional steel or non-tooth substance removing plastic curettes during supportive periodontal therapy (SPT). J Clin Periodontol. 1999 Nov;26(11):742-7. doi: 10.1034/j.1600-051x.1999.t01-6-261101.x. PMID 10589810
- [Background] Newton JT, Asimakopoulou K. Managing oral hygiene as a risk factor for periodontal disease: a systematic review of psychological approaches to behaviour change for improved plaque control in periodontal management. J Clin Periodontol. 2015 Apr;42 Suppl 16:S36-46. doi: 10.1111/jcpe.12356. PMID 25639708